## Cover Page: Consent Forms Last Updated/Approved January 13, 2019





#### Safe South Africa

Integrated Prevention of HIV Risk and Intimate Partner Violence among Adolescents in South Africa

<u>ADULT</u> Consent Form Giving <u>PERMISSION</u> for Children to Choose Participation in PROGRAM PILOT 1

Version 3 January 13, 2019

Study Implementers: South African Medical Research Council (South Africa) & Brown

University School of Public Health (USA) & Rhode Island Hospital (USA)

Study Sponsors: USA National Institute of Mental Health

**Principal Investigators:** Dr. Caroline Kuo & Dr. Catherine Mathews **Co-Investigators:** Dr. Abigail Harrison & Dr. Lindsay Orchowski

Introduction

We ask your permission to invite your child to take part in a study. Before you can make an informed decision about whether we can invite your child to take part in the study, you should understand what the study is about and the risks and benefits. This process is called informed consent. This document gives you information on what will take place in the study. The goal of this study is to find out what young people think about a new program called Safe South Africa. The program teaches young people how to become young leaders by protecting their health and the health of others. This includes discovering ways to create strong and healthy relationships, prevent violence, and promote health relating to diseases such as HIV.

## Who should provide consent?

The following adults can provide consent: (1) the *parent* (including adoptive parents); (2) if no parent, the *guardian* (either court-appointed OR as indicated by the parent in a Will); (3) if no guardian, a *foster parent*; (4) if no foster parent, a *caregiver* (any person other than a parent or guardian, who cares for a child); (5) and if the child is from a child-headed household with no supervisory adult, a *trusted adult nominated by the minor*.

## Why are we doing this study?

Young people are vulnerable to violence and sexual health problems. Teaching young people skills for preventing violence and protecting their sexual health in future relationships when they are young – before they start any risk behaviors – is the best way to protect them. We are doing this study to create a Safe South Africa program that fits the needs of young people. For the program to succeed, we need to understand what young people think of this program. This is a prevention program; this means that young people can join the study even if they have never been in a relationship, never had sex, never experienced violence, and are currently living with or without HIV.

# Study participation is voluntary.

Study participation is voluntary. This means joining the study (or NOT joining) is entirely up to the potential participant.

### What will happen in the study?

- 1. Participants complete a questionnaire that gathers background information (e.g., age, population group, language, etc.); self-reported health behaviors (e.g. any sexual experiences, HIV status, mental health, violence); and experience in relationships. This questionnaire will be repeated 1 month after the program Safe South Africa is completed, and 6 months after the program is completed. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire at the beginning, 60 Rand (consisting of 35 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire at 1 month, and 70 Rand (consisting of 45 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire at 6 months.
- 2. Participants will receive Safe South Africa. This program takes place in 2-hour sessions, once a week for a total of two weeks after school, on or near school premises. The program will take place with other teenage boys and be facilitated by our research team and includes discussion, debate, and activities where practice and gain confidence in new skills. In the program we explore ways teenage boys can become young leaders by protecting their own health and the health of others, and discover ways to create strong and healthy relationships. In the first session of the program, participants will fill out a brief assessment. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for filling out the assessment. In the second session of the program participants will fill out a brief assessment. Participants will receive 60 Rand (consisting of 35 Rand to offset time and 25 Rand to offset travel costs) for filling out the assessment.

# Risks of participating

Possible risks

We talk about sensitive topics such as violence, relationships, and health including HIV, sex, and mental health. Speaking about some of these topics can be uncomfortable. Another risk is a breach in confidentiality because of the group. Our research team will make every effort to keep personal information private and confidential but we cannot guarantee others in the group will keep information private. We will not share responses with parents (or adults in this role), teachers, or school principals. You should also be aware, however, that there are times that the law requires that we share certain information. For example South African law requires researchers and health care workers to report abuse or neglect of children. Thus, if participants talk to us about any incident of child abuse (physical abuse, sexual abuse or neglect perpetrated by a parent/guardian or caretaker), or being a victim of sexually assault or rape, we are required by law to report this information to the proper authorities to keep them safe and our team will immediately contact the study Principal Investigators (PIs), Drs. Mathews and Kuo. We will offer referrals to support organizations and report to Childline South Africa who will initiate contact with social workers and police. If participants tell us about sex between someone under 16 years (12-15 years) with a partner who is between (12-15 years), and their age is more than two years apart or between 15 or younger who is having sex with someone who is 18 years or older, we will contact the study PIs, Department of Social Development, and report to Childline with onwards reporting to social workers and/or police as necessary. We also are required by law to report if participants want to harm self or others to Childline, doctors and/or police. We advise you to consider these situations which require reporting carefully and what it means for you and your family.

How will we minimize these risks?

Paper information that we collect will be kept locked in the private offices of our study team. Other information will be kept on a computer file. Computer files will be protected by passwords that only researchers working on the project will know. Information given to us will NOT be seen by parents or teachers. Information provided will be kept for at least 5 years after the final report to study funders or after the end date of the project, whichever is later.

## **Confidentiality**

Our research team will make every effort to keep personal information private and confidential. When findings are presented from this study, any personally identifiable information (name, address, phone number) will be replaced with a unique study number. We will not share information about anything disclosed to our research team except in cases of imminent risk of harm to self or others; perpetration of rape or sexual assault with an identifiable victim; and legally mandated reporting requirements as outlined by South Africa's Children's Act including known or reasonably suspected incidents of deliberate neglect or physical, sexual, or emotional abuse of a child. If our research team is given such information, we are required to report it to the authorities such as child welfare and/or the police. These records may be reviewed by the sponsor of the study (USA National Institutes of Health and their representatives, the institutional ethics committees involved in this study, and study staff). Because we cannot guarantee others in the group will keep information private, participants should share only what they feel comfortable sharing in the group.

### **Benefits**

There may not be direct benefits from being in this study. Young people may benefit from this study later. The information gathered in study helps us design a program that can help young people stay healthy.

## What happens if you do not want to take part?

There is no penalty for choosing not to join the study or withdrawing from the study. Participants can stop taking part in the study at any time. A decision to join (or NOT join) does not affect benefits from schools, clinics, the community, or social services. If the researcher feels it is in participant's best interest, they may end study participation at any time.

# Persons to contact for problems or questions:

| • | If you have any questions | s about the stud | dy you may con | tact one of the | research | iers: |
|---|---|---|---|---|---|---|
| Se | nior researcher (TBC): Tel | • | , E-mail: _ | | | |

- If you have any questions about the study you may contact the principal investigators: Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline-kuo@brown.edu">caroline-kuo@brown.edu</a>)
- If you fall ill, suffer any side effects or if you are injured during study activities, please immediately contact:

Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline\_kuo@brown.edu">caroline\_kuo@brown.edu</a>) The SAMRC, has taken out insurance to cover you as a research participant.

• If you have any problems with the way the survey was done/concerns about your rights in the survey you may contact any one of the research ethics committees which has approved this study:

Professor Danie du Toit as chairperson who can be contacted via Adri Labuschagne- South African Medical Research Council, PO Box 19070, Tygerberg 7505, Western Cape South Africa, Tel: 021 938 0687, E-mail: <a href="mailto:adri.labuschagne@mrc.ac.za">adri.labuschagne@mrc.ac.za</a> OR Brown University Research Protections Office (Telephone: +1 401-863-3050 or toll-free at: +1 866-309-2095).

| For parent/guardian/foster parent/caregiver/trusted adult to complete: |
|---|
| I, (name and |
| surname) have had all of the above information explained and I understand the explanation. I |
| have been given answers to my questions about the study. |
| ☐ I GIVE PERMISSION for my child to decide to participate in this study and I have |
| received a copy of the information sheet. |
| ☐ I GIVE PERMISSION to be contacted for follow-up for this study and future studies. |
| □ Signature: |
| ☐ Today's date: (day)/ (month) / (year) |
| For witness to complete (if applicable): If the parent/guardian/foster parent/caregiver/trusted adult is unable to sign: Name and surname of witness: Signature of witness: Today's date: (day)/ (month) / (year) |





#### Safe South Africa

Integrated Prevention of HIV Risk and Intimate Partner Violence among Adolescents in South Africa

<u>ADULT</u> Consent Form Giving <u>PERMISSION</u> for Children to Choose Participation in <u>PILOT 2</u> SURVEY

Version 3 January 13, 2019

Study Implementers: South African Medical Research Council (South Africa) & Brown

University School of Public Health (USA) & Rhode Island Hospital (USA)

Study Sponsors: USA National Institute of Mental Health

**Principal Investigators:** Dr. Caroline Kuo & Dr. Catherine Mathews **Co-Investigators:** Dr. Abigail Harrison & Dr. Lindsay Orchowski

### Introduction

We ask your permission to invite your child to take part in a study. Before you can make an informed decision about whether we can invite your child to take part in the study, you should

<u>ADULT</u> Consent Form Giving <u>PERMISSION</u> for Children to Choose Participation in <u>PROGRAM PILOT 1</u> Version 3 January 13, 2019 understand what the study is about and the risks and benefits. This process is called informed consent. This document gives you information on what will take place in the study. The goal of this study is to find out what young people think about a new program called Safe South Africa. The program teaches young people how to become young leaders by protecting their health and the health of others. This includes discovering ways to create strong and healthy relationships, prevent violence, and promote health relating to diseases such as HIV.

# Who should provide consent?

The following adults can provide consent: (1) the *parent* (including adoptive parents); (2) if no parent, the *guardian* (either court-appointed OR as indicated by the parent in a Will); (3) if no guardian, a *foster parent*; (4) if no foster parent, a *caregiver* (any person other than a parent or guardian, who cares for a child); (5) and if the child is from a child-headed household with no supervisory adult, a *trusted adult nominated by the minor*.

### Why are we doing this study?

Young people are vulnerable to violence and sexual health problems. Teaching young people skills for preventing violence and protecting their sexual health in future relationships when they are young – before they start any risk behaviors – is the best way to protect them. We are doing this study to create a Safe South Africa program that fits the needs of young people. For the program to succeed, we need to understand what young people think of this program. This is a prevention program; this means that young people can join the study even if they have never been in a relationship, never had sex, never experienced violence, and are currently living with or without HIV.

## Study participation is voluntary.

Study participation is voluntary. This means joining the study (or NOT joining) is entirely up to the potential participant.

### What will happen in the study?

1. Participants complete a questionnaire that gathers background information (e.g., age, population group, language, etc.); self-reported health behaviors (e.g. any sexual experiences, HIV status, mental health, violence); and experience in relationships. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire.

## Risks of participating

Possible risks

We talk about sensitive topics such as violence, relationships, and health including HIV, sex, and mental health. Speaking about some of these topics can be uncomfortable. We will not share responses with parents (or adults in this role), teachers, or school principals. You should also be aware, however, that there are times that the law requires that we share certain information. For example South African law requires researchers and health care workers to report abuse or neglect of children. Thus, if participants talk to us about any incident of child abuse (physical abuse, sexual abuse or neglect perpetrated by a parent/guardian or caretaker), or being a victim of sexually assault or rape, we are required by law to report this information to the proper authorities to keep them safe and our team will immediately contact the study Principal

Investigators (PIs), Drs. Mathews and Kuo. We will offer referrals to support organizations and report to Childline South Africa who will initiate make contact with social workers and police. If participants tell us about sex between someone under 16 years (12-15 years) with a partner who is between (12-15 years), and their age is more than two years apart or between 15 or younger who is having sex with someone who is 18 years or older, we will contact the study PIs, Department of Social Development, and report to Childline with onwards reporting to social workers and/or police as necessary. We also are required by law to report if participants want to harm self or others to Childline, doctors and/or police. We advise you to consider these situations which require reporting carefully and what it means for you and your family.

### How will we minimize these risks?

Paper information that we collect will be kept locked in the private offices of our study team. Other information will be kept on a computer file. Computer files will be protected by passwords that only researchers working on the project will know. Information given to us will NOT be seen by parents or teachers. Information provided will be kept for at least 5 years after the final report to study funders or after the end date of the project, whichever is later.

## **Confidentiality**

Our research team will make every effort to keep personal information private and confidential. When findings are presented from this study, any personally identifiable information (name, address, phone number) will be replaced with a unique study number. We will not share information about anything disclosed to our research team except in cases of imminent risk of harm to self or others; perpetration of rape or sexual assault with an identifiable victim; and legally mandated reporting requirements as outlined by South Africa's Children's Act including known or reasonably suspected incidents of deliberate neglect or physical, sexual, or emotional abuse of a child. If our research team is given such information, we are required to report it to the authorities such as child welfare and/or the police. These records may be reviewed by the sponsor of the study (USA National Institutes of Health and their representatives, the institutional ethics committees involved in this study, and study staff).

### **Benefits**

There may not be direct benefits from being in this study. Young people may benefit from this study later. The information gathered in study helps us design a program that can help young people stay healthy.

## What happens if you do not want to take part?

There is no penalty for choosing not to join the study or withdrawing from the study. Participants can stop taking part in the study at any time. A decision to join (or NOT join) does not affect benefits from schools, clinics, the community, or social services. If the researcher feels it is in participant's best interest, they may end study participation at any time.

# Persons to contact for problems or questions:

• If you have any questions about the study you may contact one of the researchers:

| Senior researcher (TBC): Tel:, E-mail: |
|---|
| If you have any questions about the study you may contact the principal investigators: |
| Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, |
| Гудеrberg, 7505. Tel. 021-938 0454, E-mail: <u>cathy.mathews@mrc.ac.za</u> OR Dr. Caroline Kuo at |
| Brown University (121 South Main Street, Box G-S121-4 <sup>th</sup> Floor, Providence, Rhode Island, |
| 02912, USA; Telephone: +1 401-864-5453; Email: <u>caroline_kuo@brown.edu</u> ) |
| If you fall ill, suffer any side effects or if you are injured during study activities, please |
| immediately contact: |
| Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, |
| Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at |
| Brown University (121 South Main Street, Box G-S121-4 <sup>th</sup> Floor, Providence, Rhode Island, |
| 02912, USA; Telephone: +1 401-864-5453; Email: caroline_kuo@brown.edu) |
| The SAMRC, has taken out insurance to cover you as a research participant. |
| If you have any problems with the way the survey was done/concerns about your rights in the |
| survey you may contact any one of the research ethics committees which has approved this |
| study: |
| Professor Danie du Toit as chairperson who can be contacted via Adri Labuschagne- South |
| African Medical Research Council, PO Box 19070, Tygerberg 7505, Western Cape South |
| Africa, Tel: 021 938 0687, E-mail: adri.labuschagne@mrc.ac.za OR Brown University Research |
| Protections Office (Telephone: +1 401-863-3050 or toll-free at: +1 866-309-2095). |
| For parent/guardian/foster parent/caregiver/trusted adult to complete: |
| I, (name and |
| surname) have had all of the above information explained and I understand the explanation. I |
| have been given answers to my questions about the study. |
| ☐ I GIVE PERMISSION for my child to decide to participate in this study and I have |
| received a copy of the information sheet. |
| ☐ I GIVE PERMISSION to be contacted for follow-up for this study and future studies. |
| ☐ Signature: |
| ☐ Today's date: (day)/ (month) / (year) |
| For witness to complete (if applicable). |
| For witness to complete (if applicable): If the parent/guardian/foster parent/caregiver/trusted adult is unable to sign: |
| Name and surname of witness: |
| Signature of witness: (month) / (year) |
| today s date (day)/ (month) / (year) |





# **Safe South Africa**

Integrated Prevention of HIV Risk and Intimate Partner Violence among Adolescents in South Africa

<u>ADULT</u> Consent Form Giving <u>PERMISSION</u> for Children to Choose Participation in <u>PILOT 2</u> PROGRAM AND SURVEYS

Version 3 January 13, 2019

Study Implementers: South African Medical Research Council (South Africa) & Brown

University School of Public Health (USA) & Rhode Island Hospital (USA)

Study Sponsors: USA National Institute of Mental Health

**Principal Investigators:** Dr. Caroline Kuo & Dr. Catherine Mathews **Co-Investigators:** Dr. Abigail Harrison & Dr. Lindsay Orchowski

### Introduction

We ask your permission to invite your child to take part in a study. Before you can make an informed decision about whether we can invite your child to take part in the study, you should understand what the study is about and the risks and benefits. This process is called informed consent. This document gives you information on what will take place in the study. The goal of this study is to find out what young people think about a new program called Safe South Africa. The program teaches young people how to become young leaders by protecting their health and the health of others. This includes discovering ways to create strong and healthy relationships, prevent violence, and promote health relating to diseases such as HIV.

## Who should provide consent?

The following adults can provide consent: (1) the *parent* (including adoptive parents); (2) if no parent, the *guardian* (either court-appointed OR as indicated by the parent in a Will); (3) if no guardian, a *foster parent*; (4) if no foster parent, a *caregiver* (any person other than a parent or guardian, who cares for a child); (5) and if the child is from a child-headed household with no supervisory adult, a *trusted adult nominated by the minor*.

## Why are we doing this study?

Young people are vulnerable to violence and sexual health problems. Teaching young people skills for preventing violence and protecting their sexual health in future relationships when they are young – before they start any risk behaviors – is the best way to protect them. We are doing this study to create a Safe South Africa program that fits the needs of young people. For the program to succeed, we need to understand what young people think of this program. This is a prevention program; this means that young people can join the study even if they have never been in a relationship, never had sex, never experienced violence, and are currently living with or without HIV.

### Study participation is voluntary.

Study participation is voluntary. This means joining the study (or NOT joining) is entirely up to the potential participant.

### What will happen in the study?

Participants will be randomized to get the Safe South Africa program <u>OR</u> a package of written health information. Being randomized means being assigned to get the Safe South Africa program OR a package of written health information is entire by <u>chance</u>. Assignment to the Safe South Africa program <u>OR</u> a package of written health information <u>cannot be changed</u>.

- 1. Half of the participants in the study will be assigned to Safe South Africa. These participants will receive Safe South Africa. This program takes place in 2-hour sessions, once a week for a total of two weeks after school, on or near school premises. The program will take place with other teenage boys and be facilitated by our research team and includes discussion, debate, and activities to practice new skills for healthy lives. In the program we explore ways teenage boys can become young leaders by protecting their own health and the health of others, and discover ways to create strong and healthy relationships. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for attending the enrollment session and filling out the first session assessment. In the second session of the program participants will fill out a brief assessment. Participants will receive 60 Rand to (consisting of 35 Rand to offset time and 25 Rand to offset travel costs) for filling out the assessment.
- 2. <u>Half of the participants in the study will be assigned to receive written health information</u>. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for the enrollment session.
- 3. <u>All</u> participants complete a questionnaire that gathers background information (e.g., age, population group, language, etc.); self-reported health behaviors (e.g. any sexual experiences, HIV status, mental health, violence); and experience in relationships. This questionnaire will be repeated 1 month after the program Safe South Africa is completed, and 6 months after the program is completed. Participants will receive 60 Rand for the questionnaire at 1 month, and 70 Rand for the questionnaire at 6 months.

## Risks of participating

Possible risks

We talk about sensitive topics such as violence, relationships, and health including HIV, sex, and mental health. Speaking about some of these topics can be uncomfortable. Another risk is a breach in confidentiality because of the group. Our research team will make every effort to keep personal information private and confidential but we cannot guarantee others in the group will keep information private. We will not share responses with parents (or adults in this role), teachers, or school principals. You should also be aware, however, that there are times that the law requires that we share certain information. For example South African law requires researchers and health care workers to report abuse or neglect of children. Thus, if participants talk to us about any incident of child abuse (physical abuse, sexual abuse or neglect perpetrated by a parent/guardian or caretaker), or being a victim of sexually assault or rape, we are required by law to report this information to the proper authorities to keep them safe and our team will immediately contact the study Principal Investigators (PIs), Drs. Mathews and Kuo. We will offer referrals to support organizations and report to Childline South Africa who will initiate make contact with social workers and police. If participants tell us about sex between someone under 16 years (12-15 years) with a partner who is between (12-15 years), and their age is more than two years apart or between 15 or younger who is having sex with someone who is 18 years or older, we will contact the study PIs, Department of Social Development, and report to Childline with onwards reporting to social workers and/or police as necessary. We also are

required by law to report if participants want to harm self or others to Childline, doctors and/or police. We advise you to consider these situations which require reporting carefully and what it means for you and your family.

How will we minimize these risks?

Paper information that we collect will be kept locked in the private offices of our study team. Other information will be kept on a computer file. Computer files will be protected by passwords that only researchers working on the project will know. Information given to us will NOT be seen by parents or teachers. Information provided will be kept for at least 5 years after the final report to study funders or after the end date of the project, whichever is later.

## **Confidentiality**

Our research team will make every effort to keep personal information private and confidential. When findings are presented from this study, any personally identifiable information (name, address, phone number) will be replaced with a unique study number. We will not share information about anything disclosed to our research team except in cases of imminent risk of harm to self or others; perpetration of rape or sexual assault with an identifiable victim; and legally mandated reporting requirements as outlined by South Africa's Children's Act including known or reasonably suspected incidents of deliberate neglect or physical, sexual, or emotional abuse of a child. If our research team is given such information, we are required to report it to the authorities such as child welfare and/or the police. These records may be reviewed by the sponsor of the study (USA National Institutes of Health and their representatives, the institutional ethics committees involved in this study, and study staff). Because we cannot guarantee others in the group will keep information private, participants should share only what they feel comfortable sharing in the group.

### **Benefits**

There may not be direct benefits from being in this study. Young people may benefit from this study later. The information gathered in study helps us design a program that can help young people stay healthy.

### What happens if you do not want to take part?

There is no penalty for choosing not to join the study or withdrawing from the study. Participants can stop taking part in the study at any time. A decision to join (or NOT join) does not affect benefits from schools, clinics, the community, or social services. If the researcher feels it is in participant's best interest, they may end study participation at any time.

## Persons to contact for problems or questions:

| • | If you have any questions about the study you may contact one of the researchers: |
|---|---|
| Se | enior researcher (TBC): Tel:, E-mail: |
| • | If you have any questions about the study you may contact the principal investigators: |
| As | ssoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, |
| Ty | ygerberg, 7505. Tel. 021-938 0454, E-mail: cathy.mathews@mrc.ac.za OR Dr. Caroline Kuo at |
| Bi | rown University (121 South Main Street, Box G-S121-4th Floor, Providence, Rhode Island, |
| 02 | 2912, USA; Telephone: +1 401-864-5453; Email: caroline kuo@brown.edu) |

• If you fall ill, suffer any side effects or if you are injured during study activities, please immediately contact:

Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline\_kuo@brown.edu">caroline\_kuo@brown.edu</a>) The SAMRC, has taken out insurance to cover you as a research participant.

• If you have any problems with the way the survey was done/concerns about your rights in the survey you may contact any one of the research ethics committees which has approved this study:

Professor Danie du Toit as chairperson who can be contacted via Adri Labuschagne- South African Medical Research Council, PO Box 19070, Tygerberg 7505, Western Cape South Africa, Tel: 021 938 0687, E-mail: <a href="mailto:adri.labuschagne@mrc.ac.za">adri.labuschagne@mrc.ac.za</a> OR Brown University Research Protections Office (Telephone: +1 401-863-3050 or toll-free at: +1 866-309-2095).

| For parent/guardian/foster parent/caregiver/trusted adult to complete: |
|---|
| I, (name and |
| surname) have had all of the above information explained and I understand the explanation. I |
| have been given answers to my questions about the study. |
| ☐ I GIVE PERMISSION for my child to decide to participate in this study and I have |
| received a copy of the information sheet. |
| ☐ I GIVE PERMISSION to be contacted for follow-up for this study and future studies. |
| ☐ Signature: |
| $\square$ Today's date: (day)/ (month) / (year) |
| For witness to complete (if applicable): |
| If the parent/guardian/foster parent/caregiver/trusted adult is unable to sign: |
| Name and surname of witness: |
| Signature of witness: |
| <b>Today's date</b> : (day)/ (month) / (year) |



School of Public Health

### Safe South Africa

Integrated Prevention of HIV Risk and Intimate Partner Violence among Adolescents in South Africa

TEENAGER Assent Form for Participation in PROGRAM PILOT 1

## Version 3 January 13, 2019

Note to researcher: Only teenagers who have provided you with a written signed adult consent form can participate in the informed assent process. This signed assent form should be attached to the signed adult consent form.

Study Implementers: South African Medical Research Council (South Africa) & Brown

University School of Public Health (USA) & Rhode Island Hospital (USA)

Study Sponsors: USA National Institute of Mental Health

**Principal Investigators:** Dr. Caroline Kuo & Dr. Catherine Mathews **Co-Investigators:** Dr. Abigail Harrison & Dr. Lindsay Orchowski

Introduction

We ask you to take part in a study. Before you can make an informed decision about whether you want to take part in the study, you should understand what the study is about and the risks and benefits. This process is called informed assent. This document gives you information on what will take place in the study. The goal of this study is to find out what young people think about a new program called Safe South Africa. The program teaches young people how to become young leaders by protecting their health and the health of others. This includes discovering ways to create strong and healthy relationships, prevent violence, and promote health relating to diseases such as HIV.

# Why are we doing this study?

Young people are vulnerable to violence and sexual health problems. Teaching young people skills for preventing violence and protecting their sexual health in future relationships when they are young – before they start any risk behaviors – is the best way to protect them. We are doing this study to create a Safe South Africa program that fits the needs of young people. For the program to succeed, we need to understand what young people think of this program. This is a <u>prevention</u> program; this means that young people can join the study even if they have never been in a relationship, never had sex, never experienced violence, and are currently living with or without HIV.

### Study participation is voluntary.

Study participation is voluntary. This means joining the study (or NOT joining) is entirely up to you.

# What will happen in the study?

- 1. You complete a questionnaire that gathers background information (e.g., age, population group, language, etc.); self-reported health behaviors (e.g. any sexual experiences, HIV status, mental health, violence); and experience in relationships. This questionnaire will be repeated 1 month after the program Safe South Africa is completed, and 6 months after the program is completed. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire at the beginning, 60 Rand (consisting of 35 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire at 1 month, and 70 Rand (consisting of 45 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire at 6 months.
- 2. You will participate in Safe South Africa. This program takes place in 2-hour sessions, once a week for a total of two weeks after school, on or near school premises. The program will take place with other teenage boys and be facilitated by our research team and includes discussion, debate, and activities where you practice and gain confidence in new skills. In the program we explore ways to become a young leader by protecting your health and the health of others, and discover ways to create strong and healthy relationships. In the first session of

the program, participants will fill out a brief assessment. Participants will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for filling out the assessment. In the second session of the program participants will fill out a brief assessment. Participants will receive 60 Rand (consisting of 35 Rand to offset time and 25 Rand to offset travel costs) for filling out the assessment.

# Risks of participating

Possible risks

We talk about sensitive topics such as violence, relationships, and health including HIV, sex, and mental health. Speaking about some of these topics can be uncomfortable. Another risk is a breach in confidentiality because of the group. Our research team will make every effort to keep personal information private and confidential but we cannot guarantee others in the group will keep information private. We will not share responses with parents (or adults in this role), teachers, or school principals. You should also be aware, however, that there are times that the law requires that we share certain information. For example South African law requires researchers and health care workers to report abuse or neglect of children. Thus, if you talk to us about any incident of child abuse (physical abuse, sexual abuse or neglect perpetrated by a parent/guardian or caretaker), or being a victim of sexually assault or rape, we are required by law to report this information to the proper authorities to keep you safe and our team will immediately contact the study Principal Investigators (PIs), Drs. Mathews and Kuo. We will offer referrals to support organizations and report to Childline South Africa who will initiate contact with social workers and police. If you tell us about sex with someone who is under 12 years of age, or you are under 16 years and having sex with a partner who is between 12-15 years but are more than 2 years apart, or you are under 16 and having sex with someone who is 18 years or older, we will contact the study PIs, Department of Social Development, and report to Childline with onwards reporting to social workers and/or police as necessary. We also are required by law to report if you want to harm yourself or others to Childline, doctors and/or police. We advise you to consider these situations which require reporting carefully and what it means for you.

How will we minimize these risks?

Paper information that we collect will be kept locked in the private offices of our study team. Other information will be kept on a computer file. Computer files will be protected by passwords that only researchers working on the project will know. Information given to us will NOT be seen by parents or teachers. Information provided will be kept for at least 5 years after the final report to study funders or after the end date of the project, whichever is later.

### **Confidentiality**

Our research team will make every effort to keep personal information private and confidential. When findings are presented from this study, any personally identifiable information (name, address, phone number) will be replaced with a unique study number. We will not share information about anything disclosed to our research team except in cases of imminent risk of harm to self or others; perpetration of rape or sexual assault with an identifiable victim; and legally mandated reporting requirements as outlined by South Africa's Children's Act including known or reasonably suspected incidents of deliberate neglect or physical, sexual, or emotional abuse of a child. If our research team is given such information, we are required to report it to the authorities such as child welfare and/or the police. These records may be reviewed by the sponsor of the study (USA National Institutes of Health and their representatives, the institutional ethics committees involved in this study, and study staff). Because we cannot

guarantee others in the group will keep information private, participants should share only what they feel comfortable sharing in the group.

### **Benefits**

There may not be direct benefits from being in this study. Young people may benefit from this study later. The information gathered in study helps us design a program that can help young people stay healthy.

## What happens if you do not want to take part?

There is no penalty for choosing not to join the study or withdrawing from the study. You can stop taking part in the study at any time. A decision to join (or NOT join) does not affect benefits from schools, clinics, the community, or social services. If the researcher feels it is in your best interest they may end study participation at any time

| Persons | to | contact | for | problems | or | auestions: |
|------------|----|---------|-----|-------------|-----|------------|
| 1 01 30113 | ·· | Contact | 101 | DI ODICIIIS | VI. | questions |

| interest, they may end study participation at any time. |
|---|
| Persons to contact for problems or questions: |
| • If you have any questions about the study you may contact one of the researchers: |
| Senior researcher (TBC): Tel:, E-mail: |
| • If you have any questions about the study you may contact the principal investigators: |
| Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, |
| Tygerberg, 7505. Tel. 021-938 0454, E-mail: cathy.mathews@mrc.ac.za OR Dr. Caroline Kuo at |
| Brown University (121 South Main Street, Box G-S121-4 <sup>th</sup> Floor, Providence, Rhode Island, |
| 02912, USA; Telephone: +1 401-864-5453; Email: caroline kuo@brown.edu) |
| • If you fall ill, suffer any side effects or if you are injured during study activities, please |
| immediately contact: |
| Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, |
| Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at |
| Brown University (121 South Main Street, Box G-S121-4 <sup>th</sup> Floor, Providence, Rhode Island, |
| 02912, USA; Telephone: +1 401-864-5453; Email: caroline_kuo@brown.edu) |
| The SAMRC, has taken out insurance to cover you as a research participant. |
| • If you have any problems with the way the survey was done/concerns about your rights in the |
| survey you may contact any one of the research ethics committees which has approved this |
| study: |
| Professor Danie du Toit as chairperson who can be contacted via Adri Labuschagne- South |
| African Medical Research Council, PO Box 19070, Tygerberg 7505, Western Cape South |
| Africa, Tel: 021 938 0687, E-mail: adri.labuschagne@mrc.ac.za OR Brown University Research |
| Protections Office (Telephone: +1 401-863-3050 or toll-free at: +1 866-309-2095). |
| For participant to complete: |
| I,(name and |
| surname) have had all of the above information explained and I understand the explanation. I |
| have been given answers to my questions about the study. |
| ☐ If I am under 18 years of age, my parent/guardian/foster parent/caregiver/trusted adult |
| has given me permission to decide whether I want to participate in this study. |
| ☐ I GIVE PERMISSION to be contacted for follow-up for this study and future studies. |
| ☐ Signature of participant: |
| $\square$ Today's date: $(day)/$ (month) / (year) |

## For witness to complete (if applicable):

If the teenager is unable to sign:

| Name and surnam | ie of witness | S: | | |
|---|---|---|---|---|
| Signature of witne | ess: | | | |
| Today's date: | (day)/ | (month) / | (year) | |
| For researcher to | complete: | | | |
| I | _ | | | (researcher's name and surname) |
| declare that I have | explained th | e information giv | en in this d | ocument. I provided ample time for |
| questions and answ | ered all que | stions. | | - |
| Was a copy of this | form given t | o the participant | ? | |
| □ Yes | _ | | | |
| □ No: If no, w | hy not: | | | |
| Signature of resea | rcher: | | | |
| Today's date: | (day)/ | (month) / | (year) | - |





### Safe South Africa

Integrated Prevention of HIV Risk and Intimate Partner Violence among Adolescents in South Africa

TEENAGER Assent Form for Participation in PILOT 2 SURVEY

Version 3 January 13, 2019

Note to researcher: Only teenagers who have provided you with a written signed adult consent form can participate in the informed assent process. This signed assent form should be attached to the signed adult consent form.

Study Implementers: South African Medical Research Council (South Africa) & Brown

University School of Public Health (USA) & Rhode Island Hospital (USA)

Study Sponsors: USA National Institute of Mental Health

**Principal Investigators:** Dr. Caroline Kuo & Dr. Catherine Mathews **Co-Investigators:** Dr. Abigail Harrison & Dr. Lindsay Orchowski

## Introduction

We ask you to take part in a study. Before you can make an informed decision about whether you want to take part in the study, you should understand what the study is about and the risks and benefits. This process is called informed assent. This document gives you information on what will take place in the study. The goal of this study is to find out what young people think about a new program called Safe South Africa. The program teaches young people how to become young leaders by protecting their health and the health of others. This includes discovering ways to create strong and healthy relationships, prevent violence, and promote health relating to diseases such as HIV.

### Why are we doing this study?

Young people are vulnerable to violence and sexual health problems. Teaching young people skills for preventing violence and protecting their sexual health in future relationships when they are young – before they start any risk behaviors – is the best way to protect them. We are doing this study to create a Safe South Africa program that fits the needs of young people. For the program to succeed, we need to understand what young people think of this program. This is a <u>prevention</u> program; this means that young people can join the study even if they have never been in a relationship, never had sex, never experienced violence, and are currently living with or without HIV.

## Study participation is voluntary.

Study participation is voluntary. This means joining the study (or NOT joining) is entirely up to you.

### What will happen in the study?

1. You complete a questionnaire that gathers background information (e.g., age, population group, language, etc.); self-reported health behaviors (e.g. any sexual experiences, HIV status, mental health, violence); and experience in relationships. You will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire.

## Risks of participating

Possible risks

We talk about sensitive topics such as violence, relationships, and health including HIV, sex, and mental health. Speaking about some of these topics can be uncomfortable. We will not share responses with parents (or adults in this role), teachers, or school principals. You should also be aware, however, that there are times that the law requires that we share certain information. For example South African law requires researchers and health care workers to report abuse or neglect of children. Thus, if you talk to us about any incident of child abuse (physical abuse, sexual abuse or neglect perpetrated by a parent/guardian or caretaker), or being a victim of sexually assault or rape, we are required by law to report this information to the proper authorities to keep you safe and our team will immediately contact the study Principal Investigators (PIs), Drs. Mathews and Kuo. We will offer referrals to support organizations and report to Childline South Africa who will initiate contact with social workers and police. If you tell us about sex with someone who is under 12 years of age, or you are under 16 years and having sex with a partner who is between 12-15 years but are more than 2 years apart, or you are under 16 and having sex with someone who is 18 years or older, we will contact the study PIs, Department of Social Development, and report to Childline with onwards reporting to social workers and/or police as necessary. We also are required by law to report if you want to harm yourself or others to Childline, doctors and/or police. We advise you to consider these situations which require reporting carefully and what it means for you.

### How will we minimize these risks?

Paper information that we collect will be kept locked in the private offices of our study team. Other information will be kept on a computer file. Computer files will be protected by passwords that only researchers working on the project will know. Information given to us will NOT be

seen by parents or teachers. Information provided will be kept for at least 5 years after the final report to study funders or after the end date of the project, whichever is later.

## **Confidentiality**

Our research team will make every effort to keep personal information private and confidential. When findings are presented from this study, any personally identifiable information (name, address, phone number) will be replaced with a unique study number. We will not share information about anything disclosed to our research team except in cases of imminent risk of harm to self or others; perpetration of rape or sexual assault with an identifiable victim; and legally mandated reporting requirements as outlined by South Africa's Children's Act including known or reasonably suspected incidents of deliberate neglect or physical, sexual, or emotional abuse of a child. If our research team is given such information, we are required to report it to the authorities such as child welfare and/or the police. These records may be reviewed by the sponsor of the study (USA National Institutes of Health and their representatives, the institutional ethics committees involved in this study, and study staff).

### **Benefits**

There may not be direct benefits from being in this study. Young people may benefit from this study later. The information gathered in study helps us design a program that can help young people stay healthy.

## What happens if you do not want to take part?

There is no penalty for choosing not to join the study or withdrawing from the study. You can stop taking part in the study at any time. A decision to join (or NOT join) does not affect benefits from schools, clinics, the community, or social services. If the researcher feels it is in your best interest, they may end study participation at any time.

## Persons to contact for problems or questions:

| • | If you have any questions about | ut the study you may contact one of the researchers: |
|---|---|---|
| Se | nior researcher (TBC): Tel: | , E-mail: |
| • | If you have any questions about | ut the study you may contact the principal investigators |

- Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline\_kuo@brown.edu">caroline\_kuo@brown.edu</a>)
- If you fall ill, suffer any side effects or if you are injured during study activities, please immediately contact:

Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline\_kuo@brown.edu">caroline\_kuo@brown.edu</a>) The SAMRC, has taken out insurance to cover you as a research participant.

• If you have any problems with the way the survey was done/concerns about your rights in the survey you may contact any one of the research ethics committees which has approved this study:

Professor Danie du Toit as chairperson who can be contacted via Adri Labuschagne-South African Medical Research Council, PO Box 19070, Tygerberg 7505, Western Cape South ADULT Consent Form Giving PERMISSION for Children to Choose Participation in PROGRAM PILOT 1 Version 3 January 13, 2019
Page 17 of 21

Africa, Tel: 021 938 0687, E-mail: adri.labuschagne@mrc.ac.za OR Brown University Research Protections Office (Telephone: +1 401-863-3050 or toll-free at: +1 866-309-2095).

| For participant to complete: |
|---|
| I, (name and |
| surname) have had all of the above information explained and I understand the explanation. I |
| have been given answers to my questions about the study. |
| ☐ If I am under 18 years of age, my parent/guardian/foster parent/caregiver/trusted adul |
| has given me permission to decide whether I want to participate in this study. |
| ☐ I GIVE PERMISSION to be contacted for follow-up for this study and future studies. |
| ☐ Signature of participant: (month) / (year) |
| For witness to complete (if applicable): |
| If the teenager is unable to sign: |
| Name and surname of witness: |
| Signature of witness: |
| Signature of witness: (day)/ (month) / (year) |
| For researcher to complete: |
| I (researcher's name and surname) |
| declare that I have explained the information given in this document. I provided ample time for |
| questions and answered all questions. |
| Was a copy of this form given to the participant? |
| □ Yes |
| □ No: If no, why not: |
| Signature of researcher: |
| Signature of researcher: Today's date: (day)/ (month) / (year) |





# **Safe South Africa**

Integrated Prevention of HIV Risk and Intimate Partner Violence among Adolescents in South Africa

<u>TEENAGER</u> Assent Form for Participation in <u>PILOT 2 SURVEY</u> Version 3 January 13, 2019

Note to researcher: Only teenagers who have provided you with a written signed adult consent form can participate in the informed assent process. This signed assent form should be attached to the signed adult consent form.

Study Implementers: South African Medical Research Council (South Africa) & Brown

University School of Public Health (USA) & Rhode Island Hospital (USA)

Study Sponsors: USA National Institute of Mental Health

**Principal Investigators:** Dr. Caroline Kuo & Dr. Catherine Mathews **Co-Investigators:** Dr. Abigail Harrison & Dr. Lindsay Orchowski

### Introduction

We ask you to take part in a study. Before you can make an informed decision about whether you want to take part in the study, you should understand what the study is about and the risks and benefits. This process is called informed assent. This document gives you information on what will take place in the study. The goal of this study is to find out what young people think about a new program called Safe South Africa. The program teaches young people how to become young leaders by protecting their health and the health of others. This includes discovering ways to create strong and healthy relationships, prevent violence, and promote health relating to diseases such as HIV.

## Why are we doing this study?

Young people are vulnerable to violence and sexual health problems. Teaching young people skills for preventing violence and protecting their sexual health in future relationships when they are young – before they start any risk behaviors – is the best way to protect them. We are doing this study to create a Safe South Africa program that fits the needs of young people. For the program to succeed, we need to understand what young people think of this program. This is a prevention program; this means that young people can join the study even if they have never been in a relationship, never had sex, never experienced violence, and are currently living with or without HIV.

### Study participation is voluntary.

Study participation is voluntary. This means joining the study (or NOT joining) is entirely up to you.

## What will happen in the study?

2. You complete a questionnaire that gathers background information (e.g., age, population group, language, etc.); self-reported health behaviors (e.g. any sexual experiences, HIV status, mental health, violence); and experience in relationships. You will receive 50 Rand (consisting of 25 Rand to offset time and 25 Rand to offset travel costs) for the questionnaire.

### Risks of participating

Possible risks

We talk about sensitive topics such as violence, relationships, and health including HIV, sex, and mental health. Speaking about some of these topics can be uncomfortable. We will not share responses with parents (or adults in this role), teachers, or school principals. You should also be aware, however, that there are times that the law requires that we share certain information. For example South African law requires researchers and health care workers to report abuse or neglect of children. Thus, if you talk to us about any incident of child abuse (physical abuse, sexual abuse or neglect perpetrated by a parent/guardian or caretaker), or being a victim of sexually assault or rape, we are required by law to report this information to the proper

authorities to keep you safe and our team will immediately contact the study Principal Investigators (PIs), Drs. Mathews and Kuo. We will offer referrals to support organizations and report to Childline South Africa who will initiate contact with social workers and police. If you tell us about sex with someone who is under 12 years of age, or you are under 16 years and having sex with a partner who is between 12-15 years but are more than 2 years apart, or you are under 16 and having sex with someone who is 18 years or older, we will contact the study PIs, Department of Social Development, and report to Childline with onwards reporting to social workers and/or police as necessary. We also are required by law to report if you want to harm yourself or others to Childline, doctors and/or police. We advise you to consider these situations which require reporting carefully and what it means for you.

### How will we minimize these risks?

Paper information that we collect will be kept locked in the private offices of our study team. Other information will be kept on a computer file. Computer files will be protected by passwords that only researchers working on the project will know. Information given to us will NOT be seen by parents or teachers. Information provided will be kept for at least 5 years after the final report to study funders or after the end date of the project, whichever is later.

## **Confidentiality**

Our research team will make every effort to keep personal information private and confidential. When findings are presented from this study, any personally identifiable information (name, address, phone number) will be replaced with a unique study number. We will not share information about anything disclosed to our research team except in cases of imminent risk of harm to self or others; perpetration of rape or sexual assault with an identifiable victim; and legally mandated reporting requirements as outlined by South Africa's Children's Act including known or reasonably suspected incidents of deliberate neglect or physical, sexual, or emotional abuse of a child. If our research team is given such information, we are required to report it to the authorities such as child welfare and/or the police. These records may be reviewed by the sponsor of the study (USA National Institutes of Health and their representatives, the institutional ethics committees involved in this study, and study staff).

### **Benefits**

There may not be direct benefits from being in this study. Young people may benefit from this study later. The information gathered in study helps us design a program that can help young people stay healthy.

### What happens if you do not want to take part?

There is no penalty for choosing not to join the study or withdrawing from the study. You can stop taking part in the study at any time. A decision to join (or NOT join) does not affect benefits from schools, clinics, the community, or social services. If the researcher feels it is in your best interest, they may end study participation at any time.

# Persons to contact for problems or questions:

| • | If you have any questions al | out the study you may contact one of the researchers: |
|---|---|---|
| Sei | nior researcher (TBC): Tel: _ | , E-mail: |

• If you have any questions about the study you may contact the principal investigators:

Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline\_kuo@brown.edu">caroline\_kuo@brown.edu</a>)

• If you fall ill, suffer any side effects or if you are injured during study activities, please immediately contact:

Assoc. Prof Catherine Mathews- South African Medical Research Council, PO Box 19070, Tygerberg, 7505. Tel. 021-938 0454, E-mail: <a href="mailto:cathy.mathews@mrc.ac.za">cathy.mathews@mrc.ac.za</a> OR Dr. Caroline Kuo at Brown University (121 South Main Street, Box G-S121-4<sup>th</sup> Floor, Providence, Rhode Island, 02912, USA; Telephone: +1 401-864-5453; Email: <a href="mailto:caroline\_kuo@brown.edu">caroline\_kuo@brown.edu</a>)

The SAMRC, has taken out insurance to cover you as a research participant.

• If you have any problems with the way the survey was done/concerns about your rights in the survey you may contact any one of the research ethics committees which has approved this study:

Professor Danie du Toit as chairperson who can be contacted via Adri Labuschagne- South African Medical Research Council, PO Box 19070, Tygerberg 7505, Western Cape South Africa, Tel: 021 938 0687, E-mail: <a href="mailto:adri.labuschagne@mrc.ac.za">adri.labuschagne@mrc.ac.za</a> OR Brown University Research Protections Office (Telephone: +1 401-863-3050 or toll-free at: +1 866-309-2095).

| For participant to complete: |
|---|
| I,(name and |
| surname) have had all of the above information explained and I understand the explanation. I |
| have been given answers to my questions about the study. |
| ☐ If I am under 18 years of age, my parent/guardian/foster parent/caregiver/trusted adult |
| has given me permission to decide whether I want to participate in this study. |
| ☐ I GIVE PERMISSION to be contacted for follow-up for this study and future studies. |
| • |
| ☐ Signature of participant: (day)/ (month) / (year) |
| 1 Today 3 date (day)/ (month) / (year) |
| For witness to complete (if applicable): |
| If the teenager is unable to sign: |
| Name and surname of witness: |
| Signature of witness: |
| Today's date: (day)/ (month) / (year) |
| English to the constant |
| For researcher to complete: |
| I (researcher's name and surname) |
| declare that I have explained the information given in this document. I provided ample time for |
| questions and answered all questions. |
| Was a copy of this form given to the participant? |
| □ Yes |
| □ No: If no, why not: |
| Signature of researcher: |
| <b>Today's date:</b> (day)/ (month) / (year) |